CLINICAL TRIAL: NCT03246659
Title: Phase I Clinical Trial Using a Novel CCK-2/Gastrin Receptor-localizing Radiolabelled Peptide Probe for Personalized Diagnosis and Therapy of Patients With Progressive or Metastatic Medullary Thyroid Carcinoma
Brief Title: Radiolabelled CCK-2/Gastrin Receptor Analogue for Personalized Theranostic Strategy in Advanced MTC
Acronym: GRAN-T-MTC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paola Anna Erba (Other)
Collaborators: Jagiellonian University (Other); University Hospital Freiburg (Other); Medical University Innsbruck (Other); University Medical Centre Ljubljana (Other); NATIONAL CENTRE FOR NUCLEAR RESEARCH, Poland (Unknown); Erasmus Medical Center (Other); INRASTES, NCSR Demokritos, Athens, Greece (Unknown)
Responsible Party: Sponsor-Investigator, Paola Anna Erba, Professor, Azienda Ospedaliero, Universitaria Pisana
Organization: Azienda Ospedaliero, Universitaria Pisana (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: GRAN-T-MTC
Record Dates: First submitted 2017-07-28; First posted 2017-08-11 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Medullary Thyroid Carcinoma
Keywords: medullary thyroid carcinoma; MTC; new gastrin analog; 111In-CP04; CP04 indium; personalised diagnostics; personalised therapy; theranostics; advanced MTC; CCK-2/gastrin receptor
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1 (Experimental): 111In-CP04
  Interventions: Drug: 111In-CP04
- arm 2 (Experimental): 111In-CP04 with co-administration of gelofusine/gelaspan
  Interventions: Drug: 111In-CP04 with co-administration of gelofusine/gelaspan

INTERVENTIONS:
Drug: 111In-CP04 — Radiopharmaceutical preparation
  Other Names: 111In-CP04 (DOTA-(DGlu)6-Ala-Tyr-Gly-Trp-Met-Asp-Phe-NH2
  Arms: arm 1
Drug: 111In-CP04 with co-administration of gelofusine/gelaspan — Radiopharmaceutical preparation with co-administration of gelofusine/gelaspan
  Other Names: 111In-CP04 (DOTA-(DGlu)6-Ala-Tyr-Gly-Trp-Met-Asp-Phe-NH2
  Arms: arm 2

SUMMARY:
The study is a phase I multicentre randomized, open, parallel-arm clinical trial conducted to investigate the IMP, namely 111In-CP04.

The study consists of preclinical (to establish a clinically useful formulation for the radiolabelled peptide CP04), and a clinical step. The main objective of the clinical part of the project is to establish the safety of i.v. administration of a high peptide amount and to assess the tracer biodistribution and dosimetry in MTC and normal tissues and to determine critical organs as well as the evaluation of the potential of CCK2 receptor scintigraphy to detect cancer lesions for both low (10ug) and high (50ug) peptide amount and the decrease of kidney dose after co-administration of gelofusine /gelaspan as a nephroprotective agent. To achieve this, the following study design has been accepted: the first 4 patients will receive 2 peptide amount of CP04: low peptide amount (for diagnostic purpose) and high peptide amount (for therapeutic purpose) of CP04. If no SAE is present, the remaining pts will be randomized for 2 arms: high peptide amount of 111In-CP04 with and without gelofusine/gelaspan infusion.

It is expected that CCK-2/gastrin receptor imaging will become a valid diagnostic method for a specific non-invasive staging and follow-up of patients with MTC, and treatment of recurrent and disseminated disease will be more efficient with minimized nephro- and myelotoxicity (if 111In labelled).

DETAILED DESCRIPTION:
The main goal of the study is to expand cancer preclinical research results on the usefulness of CCK-2/gastrin receptor in clinical practice. On the basis of last few years preclinical research outcome on new biomarkers, conjugate CP04 was chosen on the basis of its good stability and affinity to CCK-2/gastrin receptor in vitro, as well as its favourable biodistribution and pharmacodynamic properties in vivo, preclinically. Within this project the tracer may get a chance to be introduced to clinical practice as a more selective and efficient tool for the diagnosis, early detection and therapy of recurrent and metastatic MTC.

Furthermore, the project may become the first step to establish a new, more effective strategy for the treatment of MTC patients leading to reduction of incidence and mortality as well as improvement of quality of life. CCK-2/gastrin receptors may become viable targets for radionuclide scintigraphy and radionuclide therapy, similarly to somatostatin receptors which have been instrumental to establish nuclear medicine efficacy in clinical practice. Achieving key project objectives (i.e. investigation of patients after administration of high peptide amount of the CCK-2/gastrin receptor labelled compound, performing complete patient peptide assessment and research nephrotoxicity in patients with or without administration for nephroprotective agent gelofusine/gelaspan), we will be able to define the exact molecular profile of an individual patient and tumour. Eventually, safe and efficacious personalized treatment will be planned using radiolabelled CCK-2/gastrin ligands of higher therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

Related to the medullary cancer of the thyroid:

1. Histologically documented medullary cancer of the thyroid.
2. Presence of more than one distant or nodal, surgically untreatable metastases confirmed with either 18F-FDG PET/CT or enhanced-CT or MRI OR
3. Doubling time (DT) of serum calcitonin level less than two years prior to study entry and negative imaging.
4. Karnofsky performance status > 50%.
5. Life expectancy of more than 6 months.

   Related to the patient:
6. Male or female patients aged >18 years without upper age limit.
7. Ability to understand and willingness to sign a written informed consent document.
8. Written informed consent obtained according to international guidelines and local laws.

Exclusion Criteria:

Related to the MTC:

1. Patients with surgically treatable medullary thyroid cancer.
2. Patients with history of second malignancy other than basal cell carcinoma of the skin.

   Related to previous or concomitant therapies :
3. Participation in any other investigational trial within 3 months of study entry.
4. Previous external beam radiation therapy within two years.
5. Organ allograft requiring immunosuppressive therapy.

   Related to the patient:
6. Pregnancy, breast-feeding.
7. Known hypersensitivity to gastrin analogues.
8. Patients with concurrent illnesses that might preclude study completion or interfere with study results.
9. Patients with bladder outflow obstruction or unmanageable urinary incontinence.
10. Clinical diagnosis of disseminated intravascular coagulation.
11. Serum creatinine >170 μmol/L, GFR < 40 mL/min
12. Known history of hypersensitivity to gelofusine /gelaspan or any other contraindications to gelofusine/gelaspan infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of CP04 | 4 months
  Safety of intravenous administration of CP04 at low peptide amount (for diagnostic purpose) and high peptide amount (for therapeutic purpose) radiolabelled with 200±10% MBq of 111In will be assessed by type, frequency, severity, timing and relation to the studied radiopharmaceutical Safety of intravenous administration of CP04 at low peptide amount (for diagnostic purpose) and high peptide amount (for therapeutic purpose) radiolabelled with 200±10% MBq of 111In will be assessed by type, frequency, severity, timing and relation to the studied radiopharmaceutical administration of adverse events and laboratory abnormalities based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Uptake of 111In-CP04 in tumor and other tissues | 72 hours from 111In-CP04 injection
  The radioactivity uptake of 111In-CP04 will be assessed in the tumor lesions and in other tissues naturally expressing CCK2 receptors, based on the planar and SPECT/CT images (expressed as the ratio of counts over the region of interest (ROI) selected over the target tissue compared to the counts over the equivalent region in patient's body which is not taking up the 111In-CP04), otherwise described as target to non target ratio T/N
Pharmacokinetics of 111In-CP04 | 72 hours from 111In-CP04 injection
  Area under the selected organs concentration versus time curve
Pharmacokinetics of 111In-CP04 | 72 hours from 111In-CP04 injection
  Area under the blood concentration versus time curve

SECONDARY OUTCOMES:
Diagnostic sensitivity/specificity of 111In-CP04 to detect cancer lesions | 3 years
  Diagnostic sensitivity/specificity of 111In-CP04 to detect cancer lesions for both diagnostic and therapeutic peptide amount by Qualitative Visual Analysis (number of patients with uptake at site of lesion, the number of lesions with abnormal tracer uptake at scintigraphy, the number and site of lesions with pathological uptake detected per verifiable organ or body region relative to those detected
Comparison of pharmacokinetic/imaging effect of low and high peptide amount | 3 years
  To evaluate the influence of a low amount of CP04 peptide on the high amount of peptide vs. the high amount of peptide alone on tumour and organ uptake
Gelofusine/gelaspan injection and CP04 kidney uptake | 3 years
  To investigate the relative decrease of kidney dose after co-administration of nephroprotective agent - gelofusine/gelaspan
Dosimetry | 72 hours from 111In-CP04 injection
  Pharmacokinetics data for the assessment of organ and tissue radiation absorbed doses..

CONTACTS AND LOCATIONS:
Overall Officials: Paola Anna Erba, Professor, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (5):
- Department of Nuclear Medicine, Innsbruck Medical University, Innsbruck, Austria
- Department of Nuclear Medicine, University Hospital Freiburg, Freiburg im Breisgau, Germany
- Erasmus University Rotterdam, Rotterdam, Netherlands
- Department of Endocrinology, Jagiellonian University Medical College, Krakow, Poland
- Department of Nuclear Medicine, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Preclinical pharmacokinetics, biodistribution, radiation dosimetry and toxicity studies required for regulatory approval of a phase I clinical trial with 111In-CP04 in medullary thyroid carcinoma patients — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4948680/
- See also: From preclinical development to clinical application: Kit formulation for radiolabelling the minigastrin analogue CP04 with In-111 for a first-in-human clinical trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4817208/